CLINICAL TRIAL: NCT05101512
Title: Assessment of the Sub-gonal Arterial Revascularization of the Lower Limbs in Critical Ischemia by Venous Allograft Stored at + 4 ° C.
Brief Title: Assessment of the Sub-gonal Arterial Revascularization of the Lower Limbs in Critical Ischemia by Venous Allograft Stored at + 4 ° C (ERAV)
Acronym: ERAV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other); Private Hospital Dijon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A02444-51
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Venous Allogeneic Transplant; Occlusive Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with critical ischemia of the lower limb (Experimental): Patient eligible and scheduled for bypass in venous allograft stored at + 4 ° C with distal anastomosis below the knee
  Interventions: Behavioral: Questionnaires on quality of life after surgery

INTERVENTIONS:
Behavioral: Questionnaires on quality of life after surgery — Patient has to answer different questionnaire about quality of life, pain, functional scores

SUMMARY:
The main objective of this study is to assess the 2-year survival with salvage of the lower limb of patients who have undergone subgonal bypass grafting by venous allograft in the treatment of Occlusive Peripheral Arterial Disease (OPAD) in critical ischemia, in the absence of usable great saphenous vein.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 (under effective contraception, hormonal contraceptive or intrauterine device, if premenopausal).
* Patient with critical ischemia of the lower limb (stage 4-5-6 according to the Rutherford classification) requiring revascularization by sub-gonal bypass
* Patient eligible and scheduled for bypass in venous allograft stored at + 4 ° C with distal anastomosis below the knee
* Patient without usable autologous great Saphenous vein
* Subject affiliated or beneficiary of a social security scheme
* Patient having received the appropriate information concerning the objectives and procedures of the study and having declared his non-objection.

Exclusion Criteria:

* Use of unscheduled allografts
* Patient requiring composite bypass in AGV + autologous venous material or prosthesis
* Patient requiring replacement of infected prostheses
* Patient with acute ischemia
* Patient with severe coagulation disorders
* Patient classified physical status score 4
* Patient participating in another clinical trial
* Potential allergy to the graft
* Protected patients: Adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Survival rate of patients at 2 years with lower limb rescue | 2 years
  survival rate of patients at 2 years with lower limb rescue (time until death or amputation - amputation free survival)

CONTACTS AND LOCATIONS:
Locations (1):
- Private Hospital of Dijon, Dijon, France